CLINICAL TRIAL: NCT01060267
Title: Effect of Intravenous Bolus Infusion of Erythromycin Prior to Endoscopy in Patients Presenting With Variceal Bleeding: A Prospective, Randomized, Double- Blind ,Placebo Controlled, Trial
Brief Title: Intravenous Erythromycin Before Endoscopy in Patients With Variceal Bleeding: A Randomized, Double-Blind Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz Medical City (Other Government)
Responsible Party: Dr. Ibrahim H Altraif, King Abdul Aziz Medical City, National Guard Health Affairs, Saudi Arabia.
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC06/019
Record Dates: First submitted 2009-12-29; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Variceal Bleeding
MeSH Terms: interventions — Erythromycin; Macrolides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythromycin (Active Comparator): The patients in erythromycin group received intravenous bolus infusion of 125 mg of erythromycin lactobionate in 50 ml of normal saline
  Interventions: Drug: Erythromycin
- Placebo Group endoscopic therapy (No Intervention): Endoscopic therapy of variceal bleeding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythromycin — The patients in erythromycin group received intravenous bolus infusion of 125 mg of erythromycin lactobionate in 50 ml of normal saline
  Other Names: Macrolide Antibiotic
  Arms: Erythromycin
Drug: Placebo — patients in placebo group 50ml of normal saline over 10 minutes, 1/2 hour before endoscopy.
  Arms: Placebo Group endoscopic therapy

SUMMARY:
Objectives:

Blood in stomach & oesophagus in patients with variceal bleeding often obscures the endoscopic view & makes endoscopic intervention difficult to perform. Erythromycin, a motilin agonist induces gastric emptying. The aim of this study was to assess the effect of Erythromycin on endoscopic visibility and its outcome.

DETAILED DESCRIPTION:
Methods:

Adult patients with liver cirrhosis or stigmata of chronic liver disease presenting with hematemesis and or melena within previous 12 hours were randomized in a double blind trial to receive either 125 mg erythromycin or placebo 30 minutes before endoscopy. The primary end points were endoscopic visibility assessed by objective scoring system & mean endoscopy duration. Secondary end points were need for repeat endoscopy and blood transfusions within 24 hours of first endoscopy , endoscopy related complications and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with liver cirrhosis or stigmata of chronic liver disease presenting with hematemesis and or melena within previous 12 hours with
* Age >18 years
* Informed consent
* Hemodynamically stable patient at the time of endoscopy after resuscitation.

Exclusion Criteria:

* Known allergy to erythromycin
* Prior gastric lavage on admission
* Current use of antiarrhythmic drugs
* Prior gastric surgery
* Previous history of cardiac arrhythmias
* Concomitant use of antihistaminic drugs with possible drug interactions with erythromycin
* Prior use of other prokinetic agents
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The primary end point was to determine the effect of erythromycin on gastric cleansing and thereby quality of endoscopic visualization, reflecting the ease with which the procedure was performed in a clear stomach. | For upto 45 minutes from start to end of endoscopy

SECONDARY OUTCOMES:
The secondary end points were; 1. the need for second look endoscopy & number of blood units transfused within 24 hours after initial endoscopy; 3. Incidence of endoscopy & drug related complications and length of hospital stay. | Five to seven days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim H Altraif, MBBS, FRCP, Principal Investigator — King Abdulaziz Medical City
Locations (1):
- King Abdul Aziz Medical City, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Altraif I, Handoo FA, Aljumah A, Alalwan A, Dafalla M, Saeed AM, Alkhormi A, Albekairy AK, Tamim H. Effect of erythromycin before endoscopy in patients presenting with variceal bleeding: a prospective, randomized, double-blind, placebo-controlled trial. Gastrointest Endosc. 2011 Feb;73(2):245-50. doi: 10.1016/j.gie.2010.09.043. Epub 2010 Dec 8. PMID 21145052